CLINICAL TRIAL: NCT00702572
Title: Phase I Study of Carboplatin, Paclitaxel, Bevacizumab and Vorinostat for Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Carboplatin, Paclitaxel, Bevacizumab and Vorinostat for Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Chandra P. Belani, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 08-004
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Phase I; Advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Phase I dose escalating scheme
  Interventions: Drug: Vorinostat, Bevacizumab, Carboplatin, Paclitaxel
- 2 (Experimental): Phase 2 will evaluate the toxicities and safety profile of the 4-drug regimen.
  Interventions: Drug: Vorinostat, Bevacizumab, Carboplatin, Paclitaxel

INTERVENTIONS:
Drug: Vorinostat, Bevacizumab, Carboplatin, Paclitaxel — This dose escalating phase will enroll sequential cohorts of 3-6 patients to be entered at the following dose levels: Level -1: Days 1-14, Vorinostat 100 mg po QD; Day 3, Bevacizumab 15 mg/kg; Carboplatin 6 AUC; Paclitaxel 175 mg/m2. Level 1: Days 1-14, Vorinostat 200 mg po QD days 1-14; Day 3, Bevacizumab 15 mg/kg; Carboplatin 6 AUC; Paclitaxel 200 mg/m2. Level 2: Days 1-14, Vorinostat 300 mg po QD days 1-14; Day 3, Bevacizumab 15 mg/kg; Carboplatin 6 AUC; Paclitaxel 200 mg/m2. Level 3: Days 1-14, Vorinostat 400 mg po QD days 1-14; Day 3, Bevacizumab 15 mg/kg; Carboplatin 6 AUC; Paclitaxel 200 mg/m2. Treatment cycles will be repeated every 3 weeks. The highest dose level which <2 out of 5 patients experience dose limiting toxicity will be defined as the recommended phase II dose.
  Other Names: SAHA
  Arms: 1
Drug: Vorinostat, Bevacizumab, Carboplatin, Paclitaxel — Once the recommended phase II dose has been established from Phase I, 12 additional patients will be treated to evaluate the toxicities and safety profile of the 4-drug regimen.
  Other Names: SAHA
  Arms: 2

SUMMARY:
The primary objective of the study is to establish the phase II recommended dose of Vorinostat when administered in combination with the regimen of carboplatin, paclitaxel and bevacizumab for patients with previously untreated advanced non-small cell lunc cancer.

DETAILED DESCRIPTION:
Since the regimen of bevacizumab, carboplatin and paclitaxel has become a standard regimen for the treatment of advanced non-squamous NSCLC, new studies in this patient population will have to include this as a reference arm. Addition of a fourth anti-cancer agent has now become the new strategy to improve the outcome for advanced non-squamous NSCLC. Since the regimen of Vorinostat, Carboplatin and Paclitaxel is already in advanced stage of development it is important to study the safety and tolerability of Vorinostat in combination with the three-drug regimen of Bevacizumab, Carboplatin and Paclitaxel. Therefore, we will evaluate Vorinostat when administered in combination with the regimen of Carboplatin, Paclitaxel and Bevacizumab for patients with previously untreated advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced non-squamous NSCLC
* No prior chemotherapy for advanced disease
* ECOG performance status 0 or 1
* Measurable disease
* Life expectancy > 3 months
* Normal bone marrow, renal and hepatic function
* Ability to take oral medications
* Willingness to sign informed consent

Exclusion Criteria:

* History of brain metastasis
* Evidence of thromboembolic phenomenon and treatment with anticoagulants
* Pregnancy
* Uncontrolled inter-current illness
* Prior therapy with Paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Establish the phase II recommended dose (P2RD) of Vorinostat when administered in combination with the regimen of carboplatin, paclitaxel and bevacizumab for patients with previously untreated advanced non-small cell lung cancer. | An average of 2 years
  Participants will be followed for survival, an expected average of two years.

SECONDARY OUTCOMES:
Evaluate safety profile of 4-drug regimen. Obtain preliminary evidence regarding anti-cancer activity of the regimen. Understand mechanistic aspects of drug effect by conducting correlative science studies on peripheral blood and archived tumor tissue. | Average of 2 years
  Participants will be followed for survival, an expected average of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P Belani, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States